CLINICAL TRIAL: NCT02182037
Title: Safety, Pharmacodynamics, and Pharmacokinetics After Single Oral Administration of 1, 5, 10, 30, 100, 200 and 400 mg BIBT 1011 BS as Drinking Solution in Healthy Subjects. An Open, Placebo-controlled, Randomised Study, Double Blind at Each Dose Level
Brief Title: Safety, Pharmacodynamics, and Pharmacokinetics of BIBT 1011 BS in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1193.1
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Healthy

ARMS (2):
- BIBT 1011 BS (Experimental)
  Interventions: Drug: Single rising doses of BIBT 1011 BS
- BIBT 1011 BS placebo (Placebo Comparator)
  Interventions: Drug: BIBT 1011 BS placebo

INTERVENTIONS:
Drug: Single rising doses of BIBT 1011 BS
  Arms: BIBT 1011 BS
Drug: BIBT 1011 BS placebo
  Arms: BIBT 1011 BS placebo

SUMMARY:
A study to assess safety, pharmacokinetics and the effect of BIBT 986 BS, given as BIBT 1011 BS, on coagulation parameters.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects as determined by results of screening
* Signed written informed consent in accordance with good clinical practice (GCP) and local legislation
* Age ≥ 18 and ≤ 45 years
* Body Mass Index ≥ 18.5 and ≤ 29.9 kg/m2

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* History or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, hormonal disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of

  * allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
  * any bleeding disorder including prolonged or habitual bleeding
  * other hematologic disease
  * cerebral bleeding (e.g. after a car accident)
  * commotio cerebri
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs which might influence the results of the trial within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (>10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 5 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* History of any familial bleeding disorder
* Thrombocytes < 150000/µl

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2001-08; Primary Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Determination of activated partial thromboplastin time (aPTT) | Pre-dose, up to 48 hours after start of treatment
Determination of international normalized ration (INR) | Pre-dose, up to 48 hours after start of treatment

SECONDARY OUTCOMES:
Determination of thrombin time (TT) | Pre-dose, up to 48 hours after start of treatment
Determination of ecarin clotting time (ECT) | Pre-dose, up to 48 hours after start of treatment
Assessment of plasma concentration time profiles of BIBT 986 BS | Pre-dose, up to 48 hours after start of treatment
Maximum concentration of BIBT 986 BS in plasma (Cmax) | Pre-dose, up to 48 hours after start of treatment
Area under the concentration time curve for BIBT 986 BS (AUC) | Pre-dose, up to 48 hours after start of treatment
Time from dosing to when the plasma concentration reaches Cmax after a single extravascular dose (tmax) | Pre-dose, up to 48 hours after start of treatment
Total mean time of residence of BIBT 986 BS- molecules in the body (MRTtot) | Pre-dose, up to 48 hours after start of treatment
Apparent volume of distribution of the analytes during the terminal phase (Vz/f) | Pre-dose, up to 48 hours after start of treatment
Terminal elimination half life of BIBT 986 BS in plasma (t1/2) | Pre-dose, up to 48 hours after start of treatment
Amount excreted over the 24 hour sampling period (Ae0-24) | Pre-dose, up to 24 hours after start of treatment
Total clearance after oral administration (CLtot/F) | Pre-dose, up to 48 hours after start of treatment
Number of patients with adverse events | Up to 17 days
Assessment of BIBT 986 BS plasma concentration- aPTT relationship | Pre-dose, up to 48 hours after start of treatment